CLINICAL TRIAL: NCT01117103
Title: A Prospective, Observational Study on the Use of Glucophage XR Therapy in the Management of Patients With Type 2 Diabetes
Brief Title: A Prospective, Observational Study to Assess and Evaluate the Use of Glucophage XR Therapy in the Management of Patients With Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Marcus Klein, Regional Medical Director, Merck Pte. Ltd Singapore, an affiliate of Merk KGaA, Darmstadt, Germany
Other Study IDs: 200039-500
Record Dates: First submitted 2010-05-03; First posted 2010-05-05 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2010-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes; Diabetes Mellitus; Glucophage; Metformin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
This was an observational, prospective, multicentric study conducted in a cohort of subjects with type 2 diabetes and prescribed with Glucophage XR therapy from hospitals or clinics in Hong Kong, Indonesia, Korea, Malaysia, Philippines and Singapore. Glucophage XR is being used in the Asia Pacific region for the treatment of subjects with type 2 diabetes. This study was designed to provide information on the day to-day experience of using Glucophage XR in the management of subjects with type 2 diabetes and its use in routine clinical practice in Asia Pacific region.

DETAILED DESCRIPTION:
Glucophage (metformin) is the standard first line therapy for subjects with type 2 diabetes mellitus (DM). The consensus statement from the American Diabetes Association and the European Association for the Study of Diabetes has recommended metformin therapy in concurrent with lifestyle intervention at diagnosis. It has been well accepted that subjects' compliance with therapy tends to decrease as the dosage frequency increases and hence the regimens should be simplified as far as possible to support good compliance with therapy. The use of an extended release formulation of metformin (Glucophage XR) supports the simplification of treatment of subjects with type 2 diabetes by allowing a once daily administration of metformin.

OBJECTIVES

Primary objective:

* To assess the tolerability of Glucophage XR therapy when used in routine clinical practice in subjects with type 2 diabetes

Secondary objective:

* To assess the effectiveness of Glucophage XR therapy on the maintenance of glycaemic control

The study does not involve any active involvement of the subjects and does not require any change from the standard medical management of the subjects. Each subject will be followed upon starting Glucophage XR therapy and until at least 12 weeks of treatment or discontinuation of treatment, whichever being earlier.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with type 2 diabetes
* Subjects who have been given Glucophage XR for the treatment of the type 2 diabetes

Exclusion Criteria:

* Subjects treated with Glucophage XR before the study initiation
* Contraindicated use of Glucophage XR based on local label
* Subjects who plan to continue on another oral anti diabetic therapy during the course of the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects diagnosed with type 2 diabetes in Asia Pacific region.
Sampling Method: Non-Probability Sample
Enrollment: 3592 (Actual)
Dates: Start 2008-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who discontinue Glucophage XR treatment prematurely (< 12 weeks) due to side effects | Baseline to post-treatment visit (after at least 12 weeks of treatment from the baseline visit)

SECONDARY OUTCOMES:
Proportion of subjects experiencing at least one gastrointestinal side effect | Baseline to post-treatment visit (after at least 12 weeks of treatment from the baseline visit) or discontinuation of treatment, whichever is earlier
Proportion of subjects remaining on Glucophage XR therapy for at least 12 weeks | Baseline to post-treatment visit (after at least 12 weeks of treatment from the baseline visit)
Incidence of side effects | Baseline to post-treatment visit (after at least 12 weeks of treatment from the baseline visit) or discontinuation of treatment, whichever is earlier
Reasons for discontinuation | At the time of discontinuation before completing the 12 weeks observation of period
Change in glycosylated haemoglobin (HbA1c) levels from baseline after 12 weeks | Baseline to post-treatment visit (after at least 12 weeks of treatment from the baseline visit)

CONTACTS AND LOCATIONS:
Overall Officials: Dr Marcus Klein, MD, PhD, Study Director — Merck Pte. Ltd., Singapore
Locations (1):
- Kevin Tan Clinic For Diabetes, Thyroid & Hormones Pte Ltd, Mount Elizabeth, Singapore